CLINICAL TRIAL: NCT04909047
Title: The Effectiveness of Parassacral Transcutaneous Stimulation Compared to Tibial Transcutaneous Stimulation, Home Protocol and Behavioral Therapy in the Treatment of Female Hyperative Bladder: Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Centro AA Pelvico
Record Dates: First submitted 2021-05-19; First posted 2021-06-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Transcutaneous Electrical Nerve Stimulation; Urgent Urinary Incontinence; Bladder Hyperactive; Women
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Parasacral transcutaneous electrostimulation outpatient (Experimental): electrostimulation device
  Interventions: Device: parassacral transcutaneous electrostimulation
- transcutaneous tibial electrostimulation outpatient (Experimental): electrostimulation device
  Interventions: Device: parassacral transcutaneous electrostimulation
- home parasacral electrostimulation (Experimental): electrostimulation device
  Interventions: Device: parassacral transcutaneous electrostimulation

INTERVENTIONS:
Device: parassacral transcutaneous electrostimulation — Use of parassacral transcutaneous electrostimulation

SUMMARY:
Introduction: The overactive bladder is a highly prevalent condition, which negatively impacts the quality of life and daily activities of women. Transcutaneous electrostimulation is currently a therapeutic alternative for urinary urgency symptoms. Although it can be applied to the sacral plexus or tibial nerve, the literature shows the effectiveness of these two modalities, in isolation, but there are few scientific studies that compare them as two therapeutic alternatives. Primary objective: to evaluate the efficacy between parascutaneous electrostimulation, tibial transcutaneous stimulation, and home protocol in the treatment of female overactive bladder. Methodology: This is a clinical trial, which will include women with a clinical complaint of overactive bladder, with or without urgency-incontinence, who will be randomized into 3 groups: transcutaneous parasacral electrostimulation (EETP), transcutaneous tibial electrostimulation (EETT) and a third group, home transcutaneous parasacral electrostimulation (EETPD), will consist of women who have financial difficulties or locomotion to attend the clinic.All groups, in the first session, will be guided to conduct behavioral therapy and will receive an educational booklet with guidelines. The equipment to be used will have a wave frequency of 10 Hz, a pulse width of 700 µs and a 20-minute session, with intensities according to the participant's tolerance. The intervention protocol of the EETP group is 30 sessions, three times a week, with an active electrode in the parasacral region. For EETT, 30 sessions will also be held, three times a week, with the electrode active in the tibial region. Participants will be captured at educational events held by the Pelvic Floor Service Center in Salvador and the metropolitan region. Participants will answer the basic anamnesis questionnaires, ICIQ-OAB, ROMA III criteria, Bristol scale, Hospital Anxiety and Depression Scale, Oswestry scale, Pittsburgh sleep quality index and Female Sexual Function Index. Then, the assessment of the bladder neck and the thickness of the bladder wall will be performed by 2D ultrasonography via suprapubic and intravaginal, following the assessment protocol described for the intervention groups. Primary outcomes: clinical improvement of symptoms, urinary frequency, episodes of urgent urinary incontinence, presence of adverse effects and constipation. Secondary outcomes: quality of life, sexual function, quality of sleep, anxiety and depression, muscle function (PERFECT and electromyography), lumbar-pelvic pain (pain intensity) and ultrasound. Participants will be followed for a minimum of 12 months to verify the long-term response, returning every 3 months. Expected results: The outpatient transcutaneous parasacral electrostimulation is expected to be superior when compared to the tibial transcutaneous electrostimulation in the resolution of the symptoms of the overactive female bladder.

ELIGIBILITY:
Inclusion Criteria:

* Women with symptoms of overactive bladder, aged 18 to 65 years.

Exclusion Criteria:

* Participants who have difficulty understanding the stages of the research, report cognitive deficit or psychiatric illness, patients with congenital orthopedic / neurological diseases, overactive bladder due to neurological impairment, presence of lower urinary tract infection, sensory deficit in the sacral or tibial region, diagnosis of chronic renal failure, patients with pacemakers and implantable cardioverter defibrillators and pregnant women.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of urinary leakage episodes | 90 days
  Clinical improvement of symptoms of urinary leakage episodes analyzed by voiding diary, urofluxometry and International Consultation on Incontinence Questionnaire Overactive Bladder (ICIQ-OAB)
Reduction in urinary frequency | 90 days
  Reduction in the number of daily urination analyzed by voiding diary , urofluxometry, 2 D ultrasonography and International Consultation on Incontinence Questionnaire Overactive Bladder (ICIQ-OAB)
Clinical improvement of constipation | 90 days
  Effort in bowel movements, stool shape, number of weekly bowel movements analyzed by Rome, Bristol criterion and 2 D ultrasonography

SECONDARY OUTCOMES:
Measuring quality of life by questionnaire | 90 days
  Will be used the King´s Health Questionnaire (KHQ)
Sexual function | 90 days
  Will be used the questionnaire of Female Sexual Function (FSFI)
Quality of sleep | 90 days
  Will be used the Pittsburgh sleep quality index (PSQI)
Anxiety and depression | 90 days
  Scale of the Hospital Anxiety and Depression Scale (HADS)
Muscle function | 90 days
  Analyze through the PERFECT test and by electromyography

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Centro de Atenção ao Assoalho Pelvico, Salvador, Estado de Bahia
  - Cebtro de Atebçao ao Assolaho Pévico- Escola Bahiana de Medicina e Saúde Pública, Salvador, Estado de Bahia
  - Centro de Atenção ao assoalho pélvico, Salvador, Estado de Bahia

REFERENCES:
- [Background] Abrams P, Andersson KE, Birder L, Brubaker L, Cardozo L, Chapple C, Cottenden A, Davila W, de Ridder D, Dmochowski R, Drake M, Dubeau C, Fry C, Hanno P, Smith JH, Herschorn S, Hosker G, Kelleher C, Koelbl H, Khoury S, Madoff R, Milsom I, Moore K, Newman D, Nitti V, Norton C, Nygaard I, Payne C, Smith A, Staskin D, Tekgul S, Thuroff J, Tubaro A, Vodusek D, Wein A, Wyndaele JJ; Members of Committees; Fourth International Consultation on Incontinence. Fourth International Consultation on Incontinence Recommendations of the International Scientific Committee: Evaluation and treatment of urinary incontinence, pelvic organ prolapse, and fecal incontinence. Neurourol Urodyn. 2010;29(1):213-40. doi: 10.1002/nau.20870. No abstract available. PMID 20025020
- [Background] Irwin DE, Kopp ZS, Agatep B, Milsom I, Abrams P. Worldwide prevalence estimates of lower urinary tract symptoms, overactive bladder, urinary incontinence and bladder outlet obstruction. BJU Int. 2011 Oct;108(7):1132-8. doi: 10.1111/j.1464-410X.2010.09993.x. Epub 2011 Jan 13. PMID 21231991
- [Background] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Background] Lucas MG, Bosch RJ, Burkhard FC, Cruz F, Madden TB, Nambiar AK, Neisius A, de Ridder DJ, Tubaro A, Turner WH, Pickard RS; European Association of Urology. EAU guidelines on surgical treatment of urinary incontinence. Eur Urol. 2012 Dec;62(6):1118-29. doi: 10.1016/j.eururo.2012.09.023. Epub 2012 Sep 17. PMID 23040204
- [Background] Gormley EA, Lightner DJ, Burgio KL, Chai TC, Clemens JQ, Culkin DJ, Das AK, Foster HE Jr, Scarpero HM, Tessier CD, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline. J Urol. 2012 Dec;188(6 Suppl):2455-63. doi: 10.1016/j.juro.2012.09.079. Epub 2012 Oct 24. PMID 23098785
- [Background] Gungor Ugurlucan F, Onal M, Aslan E, Ayyildiz Erkan H, Kizilkaya Beji N, Yalcin O. Comparison of the effects of electrical stimulation and posterior tibial nerve stimulation in the treatment of overactive bladder syndrome. Gynecol Obstet Invest. 2013;75(1):46-52. doi: 10.1159/000343756. Epub 2012 Nov 16. PMID 23171636
- [Background] Svihra J, Kurca E, Luptak J, Kliment J. Neuromodulative treatment of overactive bladder--noninvasive tibial nerve stimulation. Bratisl Lek Listy. 2002;103(12):480-3. PMID 12696778
- [Background] Scaldazza CV, Morosetti C, Giampieretti R, Lorenzetti R, Baroni M. Percutaneous tibial nerve stimulation versus electrical stimulation with pelvic floor muscle training for overactive bladder syndrome in women: results of a randomized controlled study. Int Braz J Urol. 2017 Jan-Feb;43(1):121-126. doi: 10.1590/S1677-5538.IBJU.2015.0719. PMID 28124534
- [Background] Hasan ST, Robson WA, Pridie AK, Neal DE. Transcutaneous electrical nerve stimulation and temporary S3 neuromodulation in idiopathic detrusor instability. J Urol. 1996 Jun;155(6):2005-11. PMID 8618309
- [Background] Soomro NA, Khadra MH, Robson W, Neal DE. A crossover randomized trial of transcutaneous electrical nerve stimulation and oxybutynin in patients with detrusor instability. J Urol. 2001 Jul;166(1):146-9. PMID 11435843
- [Background] Nakagawa H, Kaiho Y, Namiki S, Ishidoya S, Saito S, Arai Y. Impact of sacral surface therapeutic electrical stimulation on early recovery of urinary continence after radical retropubic prostatectomy: a pilot study. Adv Urol. 2010;2010:102751. doi: 10.1155/2010/102751. Epub 2010 Apr 29. PMID 20454700
- [Background] Barroso U Jr, Lordelo P, Lopes AA, Andrade J, Macedo A Jr, Ortiz V. Nonpharmacological treatment of lower urinary tract dysfunction using biofeedback and transcutaneous electrical stimulation: a pilot study. BJU Int. 2006 Jul;98(1):166-71. doi: 10.1111/j.1464-410X.2006.06264.x. PMID 16831163
- [Background] Lordelo P, Soares PV, Maciel I, Macedo A Jr, Barroso U Jr. Prospective study of transcutaneous parasacral electrical stimulation for overactive bladder in children: long-term results. J Urol. 2009 Dec;182(6):2900-4. doi: 10.1016/j.juro.2009.08.058. Epub 2009 Oct 28. PMID 19846164
- [Background] Lordelo P, Teles A, Veiga ML, Correia LC, Barroso U Jr. Transcutaneous electrical nerve stimulation in children with overactive bladder: a randomized clinical trial. J Urol. 2010 Aug;184(2):683-9. doi: 10.1016/j.juro.2010.03.053. Epub 2010 Jun 18. PMID 20561643
- [Background] Chu FM, Dmochowski R. Pathophysiology of overactive bladder. Am J Med. 2006 Mar;119(3 Suppl 1):3-8. doi: 10.1016/j.amjmed.2005.12.010. PMID 16483862
- [Background] Coyne KS, Sexton CC, Thompson CL, Clemens JQ, Chen CI, Bavendam T, Dmochowski R. Impact of overactive bladder on work productivity. Urology. 2012 Jul;80(1):97-103. doi: 10.1016/j.urology.2012.03.039. PMID 22748868
- [Background] Krystal AD, Preud'homme XA, Amundsen CL, Webster GD. Detrusor overactivity persisting at night and preceding nocturia in patients with overactive bladder syndrome: a nocturnal cystometrogram and polysomnogram study. J Urol. 2010 Aug;184(2):623-8. doi: 10.1016/j.juro.2010.03.148. Epub 2010 Jun 19. PMID 20639027
- [Background] Kinsey D, Pretorius S, Glover L, Alexander T. The psychological impact of overactive bladder: A systematic review. J Health Psychol. 2016 Jan;21(1):69-81. doi: 10.1177/1359105314522084. Epub 2014 Mar 2. PMID 24591118
- [Background] Ge TJ, Vetter J, Lai HH. Sleep Disturbance and Fatigue Are Associated With More Severe Urinary Incontinence and Overactive Bladder Symptoms. Urology. 2017 Nov;109:67-73. doi: 10.1016/j.urology.2017.07.039. Epub 2017 Aug 4. PMID 28826875
- [Background] Ghoniem G, Stanford E, Kenton K, Achtari C, Goldberg R, Mascarenhas T, Parekh M, Tamussino K, Tosson S, Lose G, Petri E. Evaluation and outcome measures in the treatment of female urinary stress incontinence: International Urogynecological Association (IUGA) guidelines for research and clinical practice. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Jan;19(1):5-33. doi: 10.1007/s00192-007-0495-5. Epub 2007 Nov 17. No abstract available. PMID 18026681
- [Background] Shumaker SA, Wyman JF, Uebersax JS, McClish D, Fantl JA. Health-related quality of life measures for women with urinary incontinence: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program in Women (CPW) Research Group. Qual Life Res. 1994 Oct;3(5):291-306. doi: 10.1007/BF00451721. PMID 7841963
- [Background] Coyne K, Revicki D, Hunt T, Corey R, Stewart W, Bentkover J, Kurth H, Abrams P. Psychometric validation of an overactive bladder symptom and health-related quality of life questionnaire: the OAB-q. Qual Life Res. 2002 Sep;11(6):563-74. doi: 10.1023/a:1016370925601. PMID 12206577
- [Background] Coyne KS, Matza LS, Thompson CL, Kopp ZS, Khullar V. Determining the importance of change in the overactive bladder questionnaire. J Urol. 2006 Aug;176(2):627-32; discussion 632. doi: 10.1016/j.juro.2006.03.088. PMID 16813906
- [Background] Latthe P, Middleton L, Rachaneni S, McCooty S, Daniels J, Coomarasamy A, Balogun M, Duckett J, Thakar R, Goranitis I, Roberts T, Deeks J; BUS Collaborative Group. Ultrasound bladder wall thickness and detrusor overactivity: a multicentre test accuracy study. BJOG. 2017 Aug;124(9):1422-1429. doi: 10.1111/1471-0528.14503. Epub 2017 Feb 7. PMID 28176494
- [Background] Madhuvrata P, Cody JD, Ellis G, Herbison GP, Hay-Smith EJ. Which anticholinergic drug for overactive bladder symptoms in adults. Cochrane Database Syst Rev. 2012 Jan 18;1:CD005429. doi: 10.1002/14651858.CD005429.pub2. PMID 22258963
- [Background] Peters KM, Carrico DJ, MacDiarmid SA, Wooldridge LS, Khan AU, McCoy CE, Franco N, Bennett JB. Sustained therapeutic effects of percutaneous tibial nerve stimulation: 24-month results of the STEP study. Neurourol Urodyn. 2013 Jan;32(1):24-9. doi: 10.1002/nau.22266. Epub 2012 Jun 5. PMID 22674493
- [Background] Angelo PH, de Queiroz NA, Leitao ACR, Marini G, Micussi MT. Validation of the international consultation on incontinence modular questionnaire - female lower urinary tract symptoms (ICIQ-FLUTS) into brazilian portuguese. Int Braz J Urol. 2020 Jan-Feb;46(1):53-59. doi: 10.1590/S1677-5538.IBJU.2019.0234. PMID 31851458
- [Background] Rosier PFWM, Schaefer W, Lose G, Goldman HB, Guralnick M, Eustice S, Dickinson T, Hashim H. International Continence Society Good Urodynamic Practices and Terms 2016: Urodynamics, uroflowmetry, cystometry, and pressure-flow study. Neurourol Urodyn. 2017 Jun;36(5):1243-1260. doi: 10.1002/nau.23124. Epub 2016 Dec 5. PMID 27917521
- [Background] Gezginci E, Iyigun E, Yilmaz S. Comparison of 3 Different Teaching Methods for a Behavioral Therapy Program for Female Overactive Bladder: A Randomized Controlled Trial. J Wound Ostomy Continence Nurs. 2018 Jan/Feb;45(1):68-74. doi: 10.1097/WON.0000000000000398. PMID 29300292
- [Result] Coyne KS, Sexton CC, Bell JA, Thompson CL, Dmochowski R, Bavendam T, Chen CI, Quentin Clemens J. The prevalence of lower urinary tract symptoms (LUTS) and overactive bladder (OAB) by racial/ethnic group and age: results from OAB-POLL. Neurourol Urodyn. 2013 Mar;32(3):230-7. doi: 10.1002/nau.22295. Epub 2012 Jul 27. PMID 22847394